CLINICAL TRIAL: NCT06255028
Title: The CALiPSO-1 Study: A Study of CNTY-101, a CD19-targeted CAR iNK Cell Product, in Participants With Refractory B Cell-mediated Autoimmune Diseases
Brief Title: A Study of CNTY-101 in Participants With Refractory B Cell-mediated Autoimmune Diseases
Acronym: CALiPSO-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Century Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CNTY-101-151-01; 2024-518797-13 (Other: Clinical Trial Register (CTR) Number)
Record Dates: First submitted 2024-02-05; First posted 2024-02-12 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus; Lupus Nephritis; Idiopathic Inflammatory Myopathies; Diffuse Cutaneous Systemic Sclerosis
Keywords: CAR iNK; CAR NK; Cellular therapy; Systemic Lupus Erythematosus; SLE; Induced pluripotent stem cell (iPSC); Anti-CD19 therapy; CNTY-101; Autoimmune disease; Lupus Nephritis; Lupus; Idiopathic Inflammatory Myopathies; Diffuse Cutaneous Systemic Sclerosis; IIM; DcSSc; Myositis; Polymyositis; Dermatomyositis; Anti-synthetase syndrome; Systemic sclerosis; Sclerosis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Myositis; Scleroderma, Diffuse; Autoimmune Diseases; Polymyositis; Dermatomyositis; Scleroderma, Systemic; Sclerosis | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: CNTY-101 in SLE Participants (Experimental): During Part 1 (Dose Confirmation Phase), participants with SLE will undergo lymphodepleting chemotherapy (LDC) followed by administration of CNTY-101, administered 3 times over 3 weeks, during Cycle 1 (cycle length = 28 days), alone or with supplemental human recombinant interleukin 2 (IL-2).
  After completion of Cycle 1, CNTY-101 (without preceding LDC), will be administered 3 times over 3 weeks, during Cycle 2 (cycle length = 28 days), alone or with supplemental IL-2.
  During Part 2 (Dose Expansion Phase), participants will receive treatments using the recommended phase 2 regimen (RP2R) confirmed during Part 1.
  Interventions: Biological: CNTY-101; Biological: IL-2; Drug: Lymphodepleting Chemotherapy
- Arm B: CNTY-101 in LN Participants (Experimental): During Part 1 (Dose Confirmation Phase), participants with LN will undergo LDC followed by administration of CNTY-101, administered 3 times over 3 weeks, during Cycle 1 (cycle length = 28 days), alone or with supplemental IL-2.
  After completion of Cycle 1, CNTY-101 (without preceding LDC), will be administered 3 times over 3 weeks, during Cycle 2 (cycle length = 28 days), alone or with supplemental IL-2.
  During Part 2 (Dose Expansion Phase), participants will receive treatments using the RP2R confirmed during Part 1.
  Interventions: Biological: CNTY-101; Biological: IL-2; Drug: Lymphodepleting Chemotherapy
- Arm C: CNTY-101 in IIM Participants (Experimental): During Part 1 (Dose Confirmation Phase), participants with IIM will undergo LDC followed by administration of CNTY-101, administered 3 times over 3 weeks, during Cycle 1 (cycle length = 28 days), alone or with supplemental IL-2.
  After completion of Cycle 1, CNTY-101 (without preceding LDC), will be administered 3 times over 3 weeks, during Cycle 2 (cycle length = 28 days), alone or with supplemental IL-2.
  During Part 2 (Dose Expansion Phase), participants will receive treatments using the RP2R confirmed during Part 1.
  Interventions: Biological: CNTY-101; Biological: IL-2; Drug: Lymphodepleting Chemotherapy
- Arm D: CNTY-101 in DcSSC Participants (Experimental): During Part 1 (Dose Confirmation Phase), participants with DcSSC will undergo LDC followed by administration of CNTY-101, administered 3 times over 3 weeks, during Cycle 1 (cycle length = 28 days), alone or with supplemental IL-2.
  After completion of Cycle 1, CNTY-101 (without preceding LDC), will be administered 3 times over 3 weeks, during Cycle 2 (cycle length = 28 days), alone or with supplemental IL-2.
  During Part 2 (Dose Expansion Phase), participants will receive treatments using the RP2R confirmed during Part 1.
  Interventions: Biological: CNTY-101; Biological: IL-2; Drug: Lymphodepleting Chemotherapy

INTERVENTIONS:
Biological: CNTY-101 — CNTY-101 cells for intravenous (IV) infusion
Biological: IL-2 — IL-2 subcutaneous (SC) injection
Drug: Lymphodepleting Chemotherapy — LDC as prespecified in the protocol.

SUMMARY:
CALiPSO-1 is a Phase 1, multi-centre, dose-confirmation study to evaluate the safety and efficacy of CNTY-101 in participants with refractory B cell-mediated autoimmune diseases including those with moderate to severe systemic lupus erythematosus (SLE) with or without lupus nephritis (LN), idiopathic inflammatory myopathies (IIM), and diffuse cutaneous systemic sclerosis (DcSSc).

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

1. 17 years of age and older.
2. Participants must have adequate organ function as defined in the protocol.

SLE/LN-specific Inclusion Criteria:

1. Participants must have a diagnosis of SLE according to the 2019 European League Against Rheumatism/American College of Rheumatology classification criteria for systemic lupus erythematosus for at least 6 months.
2. Participants must have current or history of elevated anti-double stranded deoxyribonucleic acid (anti-dsDNA), anti-Smith, anti-histone, and/or anti-nucleosome antibodies.

SLE-specific Inclusion Criteria:

1. Participants who have:

1. A Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score of ≥8 (including at least 4 points from non-laboratory assessments; excluding alopecia, mucosal ulcers, and fever) and at least 2 British Isles Lupus Assessment Group B (BILAG B) organ system scores and/or
2. At least one British Isles Lupus Assessment Group A (BILAG A) organ system score, including cardiac (peri- or myocarditis), respiratory (pleuritis or lung involvement), vascular and renal.

LN-specific Inclusion Criteria:

1. Participants with active, biopsy-proven, proliferative LN Class III or IV, either with or without the presence of class V, according to the 2018 revised International Society of Nephrology/Renal Pathology Society (ISN/RPS) criteria. Biopsy must be within 12 months prior to Screening or during Screening.

IIM-specific Inclusion Criteria:

1. Classification of IIM (juvenile-onset IIM may be included):

1. For Dermatomyositis (DM), meet 2017 American College of Rheumatology/European Alliance of Associations of Rheumatology (ACR/EULAR) diagnostic criteria for definite or probable DM.
2. For participants with anti-synthetase syndrome (ASyS), meet Classification Criteria for anti-synthetase syndrome per the Classification Criteria for Anti-Synthetase Syndrome (CLASS) Project with a positive tRNA synthetase autoantibody at Screening or per medical history.
3. For Polymyositis (PM)/ necrotizing myopathy (NM), meet 2017 ACR/ EULAR classification criteria for definite or probable PM/NM and meet one of the following criteria:

i. Positive myositis specific antibody (MSA) at Screening or per medical history or ii. Muscle biopsy at Screening or per medical history available for review

DcSSc-specific Inclusion Criteria:

1. Meets the 2013 ACR/EULAR criteria for SSc with a total score of ≥9.
2. Meets criteria for DcSSc, including skin involvement proximal to the elbow and/or knee.
3. mRSS units ≥15 at Screening; for participants agreeing to biopsy, skin thickening from SSc in the forearm suitable for biopsy.

Exclusion Criteria:

General Exclusion Criteria:

1. Participants on hemodialysis.
2. Other comorbid conditions as defined in the protocol.
3. History of allogeneic bone marrow/hematopoietic stem cell or solid organ transplant at any time. History of autologous stem cell transplant >100 days prior to Screening is allowed.
4. Recent or clinically significant central nervous system (CNS) disease, including but not limited to cerebrovascular accident, epilepsy, severe brain injury, dementia, Parkinson's disease, cerebellar disease, seizures, organic brain syndrome, lupus headache, or psychosis at any time prior to study.
5. Thromboembolic events within last 12 months.
6. Participants with severe hepatic dysfunction, defined as grade C-Child-Pugh.

SLE-specific Exclusion Criteria:

1. Participants with BILAG A for neuropsychiatric SLE.
2. Any current, acute, and severe lupus-related flare that needs immediate treatment.
3. Drug-induced SLE rather than idiopathic SLE.
4. Participants with a diagnosis of LN Classes III, IV, V, or VI on the most current biopsy according to the 2018 revised ISN/RPS criteria.
5. Participants with estimated glomerular filtration rate (eGFR) <45 milliliters per minute per 1.73 square meter (mL/min/1.73 m^2) (measured by Chronic Kidney Disease Epidemiology Collaboration Creatinine Equation) or serum creatinine >2.5 milligrams per deciliter (mg/dL).

LN-specific Exclusion Criteria:

1. Participants with BILAG A for neuropsychiatric SLE.
2. Any severe lupus-related flare such as acute CNS lupus (eg, psychosis, seizure), catastrophic antiphospholipid syndrome, or rapidly progressive glomerulonephritis that, in the opinion of the Investigator, would cause an unacceptable safety risk.
3. Drug-induced SLE rather than idiopathic SLE.
4. Participants with predominantly LN Class V, or Class VI on the most recent biopsy according to the 2018 revised ISN/RPS criteria.
5. Participants with estimated glomerular filtration rate <30 mL/min/1.73 m^2 (measured by Chronic Kidney Disease Epidemiology Collaboration Creatinine Equation) or serum creatinine >2.5 mg/dL.

IIM- specific Exclusion Criteria:

1. Participants on hemodialysis or estimated glomerular filtration rate <45 mL/min/1.73 m^2 (measured by Chronic Kidney Disease Epidemiology Collaboration Creatinine Equation) or serum creatinine >2.5 mg/dL.
2. Have severe muscle damage as defined in the protocol.
3. Participants with ILD will be excluded if there is severe end stage lung disease as defined in the protocol.

DcSSc-specific Exclusion Criteria

1. Participants on hemodialysis or estimated glomerular filtration rate <45 mL/min/1.73 m^2 (measured by Chronic Kidney Disease Epidemiology Collaboration Creatinine Equation) or serum creatinine >2.5 mg/dL.
2. Participants with ILD will be excluded if there is severe end stage lung disease as defined in the protocol.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2025-02-06 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) and Severity of TEAEs | Up to 29 days
Percentage of Participants With Dose Limiting Toxicities (DLTs) | Up to 28 days after first CNTY-101 infusion
Recommended Phase 2 Regimen (RP2R) of CNTY-101 With/Without IL-2 (With or Without Optimized LDC) | Up to 3 months after the first CNTY-101 infusion

SECONDARY OUTCOMES:
Percentage of Participants With TEAEs and Serious Adverse Events (SAEs) | Day 1 up to 1 year
Percentage of Participants With Clinically Significant Laboratory Abnormalities and Severity of Laboratory Abnormalities | Day 1 up to 1 year
Percentage of Participants With Cytokine Release Syndrome (CRS) and Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) and Severity of CRS and ICANS | Day 1 up to 1 year
Percentage of Participants With SLE - Responder Index 4 (SRI-4) Response | Up to 1 year
Percentage of Participants With Low Disease Activity by Lupus Low Disease Activity State (LLDAS) | Up to 1 year
Percentage of Participants in Remission as Measured by Definitions of Remission in SLE (DORIS) Remission | Up to 1 year
Percentage of Participants With Total Improvement Score (TIS) ≥20, ≥40, and ≥60 | Up to 1 year
Mean TIS | Baseline up to 1 year
Change From Baseline in Each Core Set Measures (CSM) | Baseline up to 1 year
Change From Baseline in CSM Component of Manual Muscle Testing (MMT)-8 Score | Baseline up to 1 year
Change From Baseline in CSM Component of Patient Global Assessment (PtGA) | Baseline up to 1 year
Change From Baseline in CSM Component of Physician Global Assessment (PhGA) | Baseline up to 1 year
Change From Baseline in CSM Component of Muscle Enzyme Levels | Baseline up to 1 year
Change From Baseline in CSM Component of Health Assessment Questionnaire- Disability Index (HAQ-DI) Score | Baseline up to 1 year
Change From Baseline in CSM Component of Extramuscular Assessment by Myositis Disease Activity Assessment Tool (MDAAT) | Baseline up to 1 year
For Participants With Interstitial Lung Disease (ILD): Time to Improvement in Forced Vital Capacity (FVC%) ≥10% | Up to 1 year
For Participants With ILD: Percentage of Participants With Improvement in FVC% ≥10% | Up to 1 year
For Participants with ILD: Change From Baseline in Percent FVC (%FVC) | Baseline up to 1 year
For Participants With ILD: Change From Baseline in Percent Diffusion Capacity of The Lung for Carbon Monoxide (%DLCO) | Baseline up to 1 year
For Participants With ILD: Time to Progression in Interstitial Lung Disease (ILD) | Up to 1 year
For Participants With ILD: Percentage of Participants With Progression in ILD | Up to 1 year
For Participants With ILD: Change in Participant Reported Dyspnea Over Time as Measured by University of California San Diego Shortness of Breath Questionnaire (UCSD SOBQ) | Up to 1 year
Change in American College of Rheumatology Combined Response in Diffuse Cutaneous Systemic Sclerosis (ACR-CRISS) Scores | Up to 1 year
Percentage of Responders as Measured by ACR-CRISS Score | Up to 1 year
Change From Baseline in ACR-CRISS Scores | Baseline up to 1 year
Change From Baseline in Fibrosing Skin Disease Based on Modified Rodnan Skin Score (mRSS) | Baseline up to 1 year
Change From Baseline in Scleroderma Health Assessment Questionnaire (SHAQ) | Baseline up to 1 year

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Keck School of Medicine of University of Southern California, Los Angeles, California
  - UC Davis, Sacramento, California
  - Lurie Children's; Northwestern Medicine - Northwestern Medical Group, Chicago, Illinois
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Fred Hutch, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No